CLINICAL TRIAL: NCT05407064
Title: A Phase 2, Multi-center, Randomized, Double-Blind, Parallel-Group, Dose-Finding Study to Assess the Effect of Four Doses of MM-120 (LSD D-Tartrate) for the Treatment of Anxiety Symptoms
Brief Title: A Dose-Finding Study of MM-120 (LSD D-Tartrate) for the Treatment of Anxiety Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Definium Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMED008
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Generalized
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1- Placebo (Placebo Comparator): A substance that is designed to have no therapeutic value.
  Interventions: Other: Placebo
- Arm 2- 25 μg MM-120 (LSD D-Tartrate) (Experimental): A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A).
  Interventions: Drug: MM-120 (LSD D-Tartrate)
- Arm 3- 50 μg MM-120 (LSD D-Tartrate) (Experimental): A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A).
  Interventions: Drug: MM-120 (LSD D-Tartrate)
- Arm 4- 100 μg MM-120 (LSD D-Tartrate) (Experimental): A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A).
  Interventions: Drug: MM-120 (LSD D-Tartrate)
- Arm 5- 200 μg MM-120 (LSD D-Tartrate) (Experimental): A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A).
  Interventions: Drug: MM-120 (LSD D-Tartrate)

INTERVENTIONS:
Drug: MM-120 (LSD D-Tartrate) — A psychoactive substance that mediates effects mainly through an agonist activity in the serotonin 2A receptor (5-HT2A).
  Arms: Arm 2- 25 μg MM-120 (LSD D-Tartrate); Arm 3- 50 μg MM-120 (LSD D-Tartrate); Arm 4- 100 μg MM-120 (LSD D-Tartrate); Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Other: Placebo — A substance that is designed to have no therapeutic value.
  Arms: Arm 1- Placebo

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, parallel-group, dose-finding study to assess the effect of 4 doses of MM-120 (25, 50, 100 or 200 μg freebase-equivalent) for the treatment of anxiety symptoms in subjects diagnosed with generalized anxiety disorder (GAD).

DETAILED DESCRIPTION:
The study will enroll approximately 200 male and female subjects 18 years to < 75 years of age who meet DSM-5 criteria for GAD and have a minimum HAM-A Total Score of 20. Subjects on contraindicated concomitant medications, supplements or other therapeutics at Screening (Visit 1) will undergo a medication taper prior to advancing to Baseline (Visit 2).

ELIGIBILITY:
Inclusion Criteria:

* Bodyweight of ≥ 50 kg
* Body mass index [BMI] ≥ 18 to ≤ 38 mg/kg2
* Diagnosis of DSM-5 generalized anxiety disorder
* Acceptable overall medical condition to be safely enrolled into and to complete the study
* Ability to swallow capsules
* Ability to provide informed consent

Exclusion Criteria:

* Women of childbearing potential (WOCBP) (i.e., physiologically capable of becoming pregnant) who are unwilling or unable to use a highly effective method of contraception for the duration of the study, OR Men physiologically capable of fathering a child who are sexually active with WOCBP but are unwilling or unable to use barrier contraception (e.g., condom with or without spermicidal cream or jelly) for the duration of the study
* Women who are currently pregnant or breastfeeding or plan to become pregnant or breastfeed during the study
* Men who plan to donate sperm during the study
* Prior history (lifetime diagnosis) with a lifetime diagnosis of schizophrenia spectrum, or other psychotic disorders or bipolar disorder
* Has a significant risk of suicide attempt based upon medical history or has active suicidal ideation
* Unwillingness or inability to discontinue prohibited concomitant medications, supplements or other therapeutics (prescription or over-the-counter)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Preferred Research Partners, Little Rock, Arkansas
  - Irvine Center for Clinical Research, Irvine, California
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - Mountain View Clinical Research, Denver, Colorado
  - Wholeness Center, Fort Collins, Colorado
  - Segal Trials, Lauderhill, Florida
  - CNS Healthcare - Orlando, Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Uptown Research, Chicago, Illinois
  - Sunstone Therapies, Rockville, Maryland
  - SISU, Springfield, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Hassman Research Institute, Berlin, New Jersey
  - GMI - Princeton Medical Institute, Princeton, New Jersey
  - Lutheran Hospital - Cleveland Clinic, Cleveland, Ohio
  - BioBehavioral Research of Austin, Austin, Texas
  - University of Texas Health Houston, Houston, Texas
  - Cedar Clinical Research, Draper, Utah
  - Cedar Clinical Research - Murray, Murray, Utah
  - Woodstock Research Center, Woodstock, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robison R, Barrow R, Conant C, Foster E, Freedman JM, Jacobsen PL, Jemison J, Karas SM, Karlin DR, Solomon TM, Halperin Wernli M, Fava M. Single Treatment With MM120 (Lysergide) in Generalized Anxiety Disorder: A Randomized Clinical Trial. JAMA. 2025 Oct 21;334(15):1358-1372. doi: 10.1001/jama.2025.13481. PMID 40906494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 554 potential participants were screened and 356 were excluded. Of the 198 participants randomized to study treatment, 147 (74.2%) completed the study.
Period: Overall Study
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Started | 39 | 39 | 40 | 40 | 40
Completed | 26 | 29 | 29 | 33 | 30
Not Completed | 13 | 10 | 11 | 7 | 10

BASELINE CHARACTERISTICS:
Population: There were 198 participants in the Randomized Set and 198 participants in the Safety Set. Of these, 194 (98.0%) of participants were included in the Full Analysis Set and 183 (92.4%) were included in the Per Protocol Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate) | Total
Number analyzed (Participants) | 39 | 39 | 36 | 40 | 40 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.66) | 38.0 (12.08) | 45.3 (14.23) | 42.7 (14.79) | 42.1 (13.53) | 41.3 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 20 | 16 | 28 | 110
  Male | 13 | 19 | 16 | 24 | 12 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 3 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 2 | 1 | 3 | 15
  White | 30 | 33 | 29 | 36 | 33 | 161
  More than one race | 0 | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 36 | 40 | 40 | 194
Baseline HAM-A Total Score [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale (HAM-A) consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
  units on a scale | 30.3 (6.56) | 30.2 (6.05) | 30.3 (5.71) | 29.3 (6.42) | 31.0 (6.98) | 30.1 (6.44)
Baseline MADRS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Åsberg Depression Rating Scale (MADRS) - used to assess depression severity and to detect changes due to treatment. Questionnaire included 10 clinician-completed items. Each of 10 questions scored with a range of 0-6 points. An item score of 0 indicated item not present or normal, while an item score of 6 indicated severe or continuous presence of the symptoms. The total possible score was 60, and higher scores represented a more severe condition. A decrease in score by ≥ 50% indicated a response to treatment, and an actual score of ≤ 10 indicated a remission of symptoms.
  units on a scale | 27.6 (9.69) | 25.4 (7.58) | 27.7 (8.30) | 26.5 (7.99) | 28.9 (8.31) | 27.2 (8.50)
Baseline PSQL Global Score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality and disturbances over the preceding month. The questionnaire had a Component Score for each of these with a range of 0-3 points: Subjective sleep quality, Sleep latency, Sleep duration, Habitual sleep efficiency, Sleep disturbance, Use of sleeping medication, and Daytime dysfunction. The sum of the Component Scores = a Global Score (range of 0-21 points). Global Score of 0 indicated no difficulty and a Global Score of 21 indicated severe difficulty in all areas. Population: PSQL not collected in 1 participant
  units on a scale
    number analyzed (Participants) | 38 | 39 | 36 | 40 | 40 | 193
    (all) | 10.9 (4.15) | 10.7 (3.40) | 11.1 (3.43) | 11.0 (3.47) | 10.1 (3.33) | 10.8 (3.59)
Baseline CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity (CGI-S) was used to assess the subject's current severity of illness at the time of the assessment relative to the clinician's past experience with patients who have the same diagnosis. The CGI-S comprises 1 Investigator-completed (or trained rater-completed) item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness.
  units on a scale | 4.9 (0.61) | 4.9 (0.75) | 4.9 (0.62) | 4.8 (0.75) | 5.1 (0.73) | 4.9 (0.70)
Baseline PGI-S [Mean (Standard Deviation); unit: units on a scale] — The Patient Global Impression - Severity (PGI-S) is the patient-reported outcome counterpart to the CGI scale. The PGI is adapted to the patient population and can be used to measure disease severity (PGI-S). The PGI-S comprises 1 subject-completed item with 5 possible ratings (1-5). A higher score indicates more severe illness.
  units on a scale | 3.7 (0.58) | 3.8 (0.63) | 3.8 (0.62) | 3.7 (0.66) | 3.7 (0.72) | 3.8 (0.65)
Baseline SDS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) is a composite of 3 self-rated items designed to measure the extent to which 3 major domains in the patient's life (work, social life/leisure activities and family life/home responsibilities) are functionally impaired by psychiatric or medical symptoms. Total score 0-30 (0 unimpaired, 30 highly impaired). Work/school (0-10); Social life (0-10); Family life/home responsibilities (0-10).
  units on a scale | 18.9 (4.08) | 18.7 (5.10) | 17.6 (5.60) | 19.2 (5.25) | 19.9 (5.44) | 19.0 (5.19)
Baseline ASEX Female [Mean (Standard Deviation); unit: units on a scale] — The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction. Population: assessed in females only in this section.
  units on a scale
    number analyzed (Participants) | 26 | 20 | 20 | 15 | 28 | 109
    (all) | 15.7 (4.78) | 15.1 (3.41) | 16.6 (4.51) | 14.9 (4.67) | 16.6 (3.71) | 15.8 (4.25)
Baseline ASEX Male [Mean (Standard Deviation); unit: units on a scale] — The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction. Population: Males only in this section.
  units on a scale
    number analyzed (Participants) | 13 | 19 | 16 | 24 | 12 | 84
    (all) | 11.8 (3.48) | 14.2 (3.52) | 13.8 (4.18) | 12.8 (3.87) | 13.6 (5.85) | 13.2 (4.27)
Baseline ASEX with Dysfunction Female [Count of Participants; unit: Participants] — The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction. Population: Females only in this section.
  Participants
    number analyzed (Participants) | 26 | 20 | 20 | 15 | 28 | 109
    (all) | 13 | 16 | 15 | 12 | 16 | 72
Baseline ASEX with Dysfunction Male [Count of Participants; unit: Participants] — The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction. Population: Males only in this section
  Participants
    number analyzed (Participants) | 13 | 19 | 16 | 24 | 12 | 84
    (all) | 2 | 8 | 7 | 7 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Dose Response
Description: To investigate the dose-response relationship for different doses of MM120 versus placebo in change from Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Week 4. The HAM-A consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). The central rater assessed the extent to which the subject displayed each given criterion and gave a rating on a scale of 0-4, where 4 represents the most severe symptoms. Minimum score = 0, maximum score = 56. Scores are summed and the greater the total score, the more severe illness.
Time Frame: 4 weeks
Population: Full Analysis Set (FAS) All subjects in the randomized set with a valid Baseline HAM-A assessment and at least one valid post-baseline HAM-A assessment. Subjects were analyzed according to the treatment assigned. Missing data for the primary endpoint were imputed using a multiple imputation approach assuming that the missingness mechanism can be retrieved from observed data. The imputation model included the treatment group and the longitudinal sequence of HAM-A Total Score.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 39 | 39 | 40 | 40 | 40
units on a scale
  Mean Change from Baseline to Week 4 in HAM-A total score Model Averaging Method | -14.23 [-17.83 to -10.63] | -15.35 [-17.62 to -13.09] | -16.05 [-19.40 to -12.71] | -19.22 [-21.73 to -16.70] | -20.09 [-22.87 to -17.31]
  Mean Difference in HAM-A total score from Placebo | 0.0 [0.0 to 0.0] | -1.24 [-6.01 to 3.53] | -1.82 [-7.65 to 4.00] | -5.02 [-9.60 to -0.44] | -5.95 [-9.84 to -2.06]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate) vs Arm 3- 50 μg MM-120 (LSD D-Tartrate) vs Arm 4- 100 μg MM-120 (LSD D-Tartrate) vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); The primary endpoint was evaluated by determining if there was a dose-response relationship between the change from baseline to Week 4 in total HAM-A score and the dose administered using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed, and multiple comparison techniques were used to choose the model(s) likely to present the true underlying dose-response curve; Test type: Superiority — Mean change from baseline and mean difference between MM120 dose groups and placebo were estimated using model averaging method (of 3 models). The minimally efficacious dose was defined as a placebo-adjusted improvement of 2.5 points on the HAM-A, with a statistical significance set at an alpha level of 0.05; A test statistic was derived from the data using an ANCOVA model with change from Baseline to Week 4 for the HAM-A Total Score as a response variable, treatment arm and Baseline value of HAM-A Total Score as covariates. The ANCOVA model was repeated for each imputed dataset, which resulted in a set of LS mean estimates for all dose groups and the related covariance matrices. Rubin's rule was used to combine the multiple sets of LS mean estimates and the related covariance matrices to a single set of LS mean estimates of change from Baseline to Week 4 for HAM-A Total Score for all dose groups and the related covariance matrix. The SAS procedure PROC MIANALYZE was used to combine the results from imputed datasets

2. Secondary Outcome: Dose Response
Description: To investigate the dose-response relationship for different doses of MM120 versus placebo in change from Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Week 8. The HAM-A consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). The central rater assessed the extent to which the subject displayed each given criterion and gave a rating on a scale of 0-4, where 4 represents the most severe symptoms. Minimum score = 0, maximum score = 56. Scores are summed and the greater the total score, the more severe illness.
Time Frame: 8 weeks
Population: Full Analysis Set (FAS) All subjects in the randomized set with a valid Baseline HAM-A assessment and at least one valid post-baseline HAM-A assessment. Subjects were analyzed according to the treatment assigned. Missing data for key secondary endpoint were imputed using a multiple imputation approach assuming that the missingness mechanism can be retrieved from observed data. The imputation model included the treatment group and the longitudinal sequence of HAM-A Total Score.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 39 | 39 | 40 | 40 | 40
units on a scale
  Mean change from Baseline to Week 8 HAM-A total score from Model Averaging Method | -15.51 [-17.79 to -13.23] | -16.24 [-18.12 to -14.36] | -16.90 [-18.70 to -15.09] | -18.39 [-20.17 to -16.61] | -20.94 [-23.92 to -17.95]
  Mean difference from Placebo at Week 8 | 0.0 [0 to 0] | -0.76 [-1.72 to 0.20] | -1.44 [-3.08 to 0.20] | -2.92 [-5.37 to -0.46] | -5.43 [-9.46 to -1.39]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate) vs Arm 3- 50 μg MM-120 (LSD D-Tartrate) vs Arm 4- 100 μg MM-120 (LSD D-Tartrate) vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); The primary endpoint was evaluated by determining if there was a dose-response relationship between the change from baseline to Week 8 in total HAM-A score and the dose administered using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed, and multiple comparison techniques were used to choose the model(s) likely to present the true underlying dose-response curve; Test type: Superiority — [test comment as in outcome 1, analysis 1]; A test statistic was derived from the data using an ANCOVA model with change from Baseline to Week 8 for the HAM-A Total Score as a response variable, treatment arm and Baseline value of HAM-A Total Score as covariates. The ANCOVA model was repeated for each imputed dataset, which resulted in a set of LS mean estimates for all dose groups and the related covariance matrices. Rubin's rule was used to combine the multiple sets of LS mean estimates and the related covariance matrices to a single set of LS mean estimates of change from Baseline to Week 8 for HAM-A Total Score for all dose groups and the related covariance matrix. The SAS procedure PROC MIANALYZE was used to combine the results from imputed datasets

3. Secondary Outcome: Change From Baseline in HAM-A Total Score
Description: To determine the change from Baseline of 4 doses of MM120 (25, 50, 100 or 200 μg free base equivalent) compared to Placebo as measured by the change in HAM-A Total Score from Baseline to Week 4 Hamilton Anxiety Rating Scale (HAM-A) consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). The central rater assessed the extent to which the subject displayed each given criterion and gave a rating on a scale of 0-4, where 4 represents the most severe symptoms. Minimum score = 0, maximum score = 56. Scores are summed and the greater the total score, the more severe illness. Data shown are change in HAM-A Total Score from Baseline to Week 4
Time Frame: 4 weeks
Population: All randomized subjects with a valid Baseline HAM-A assessment and at least one valid post-baseline HAM-A assessment were included in the FAS. Subjects were analyzed according to the treatment assigned. Missing data was not imputed for analysis of non-key secondary efficacy endpoints or safety endpoints. No adjustment for multiplicity was performed for testing the non-key secondary and exploratory endpoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 30 | 34 | 35 | 39 | 39
units on a scale | -13.6 (9.79) | -17.2 (10.53) | -14.8 (9.96) | -20.9 (9.72) | -19.7 (9.48)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.1157, ANCOVA
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.6630, ANCOVA
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0004, ANCOVA
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0100, ANCOVA

4. Secondary Outcome: Change From Baseline in HAM-A Total Scores
Description: To determine the change from Baseline in HAM-A total scores of 4 doses of MM120 (25, 50, 100 or 200 μg free base equivalent) compared with placebo from Baseline to Week 8. Hamilton Anxiety Rating Scale (HAM-A) consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). The central rater assessed the extent to which the subject displayed each given criterion and gave a rating on a scale of 0-4, where 4 represents the most severe symptoms. Minimum score = 0, maximum score = 56. Scores are summed and the greater the total score, the more severe illness. Data shown are change in HAM-A Total Score from Baseline to Week 8
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 36 | 33
units on a scale | -15.4 (9.72) | -18.6 (10.91) | -14.5 (10.15) | -19.4 (10.28) | -21.1 (10.37)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.2309, ANCOVA
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.7218, ANCOVA
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0637, ANCOVA
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0216, ANCOVA

5. Secondary Outcome: Change From Baseline in HAM-A Total Scores
Description: To determine the change from Baseline in HAM-A total scores of 4 doses of MM120 (25, 50, 100 or 200 μg free base equivalent) compared with placebo from Baseline to End of Study (Week 12). Hamilton Anxiety Rating Scale (HAM-A) consists of the following 14 items that encompass both psychological and somatic symptoms of anxiety: Anxious mood, Tension, Fears, Insomnia, Intellectual, Depressed mood, Somatic (muscular), Somatic (sensory), Cardiovascular symptoms, Respiratory symptoms, Gastrointestinal symptoms, Genitourinary symptoms, Autonomic symptoms, and Behavior at interview (general). The central rater assessed the extent to which the subject displayed each given criterion and gave a rating on a scale of 0-4, where 4 represents the most severe symptoms. Minimum score = 0, maximum score = 56. Scores are summed and the greater the total score, the more severe illness. Data shown are change in HAM-A Total Score from Baseline to end of study (12 weeks)
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale | -14.3 (11.95) | -18.7 (10.85) | -17.3 (10.71) | -21.1 (10.35) | -22.0 (11.85)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate) vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.1006, ANCOVA
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.2225, ANCOVA
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0025, ANCOVA
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Change from Baseline: ANCOVA determination of Least Squares (LS) Mean and difference in LS Mean from placebo; Test type: Superiority; p = 0.0042, ANCOVA

6. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in depressive symptoms as measured by the MADRS. The Montgomery-Åsberg Depression Rating Scale (MADRS) - used to assess depression severity and to detect changes due to treatment. Questionnaire included 10 clinician-completed items. Each of 10 questions scored with a range of 0-6 points. An item score of 0 indicated item not present or normal, while an item score of 6 indicated severe or continuous presence of the symptoms. The total possible score was 60, and higher scores represented a more severe condition. A decrease in score by ≥ 50% indicated a response to treatment, and an actual score of ≤ 10 indicated a remission of symptoms.
Time Frame: Week 1
Population: All randomized subjects with a valid Baseline HAM-A assessment and at least one valid post-baseline HAM-A assessment were included in the FAS. Subjects were analyzed according to the treatment assigned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 33 | 38 | 36 | 38 | 36
units on a scale | -11.0 (11.62) | -12.3 (10.45) | -11.1 (10.59) | -17.6 (11.21) | -17.4 (10.66)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Change from baseline in total MADRS scores determined by the difference in means and difference between treatment and placebo (p-value determined from two-sample t-test); Test type: Superiority; p = 0.6258, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.95, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0174, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0206, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in depressive symptoms measured via the MADRS. The Montgomery-Åsberg Depression Rating Scale (MADRS) - used to assess depression severity and to detect changes due to treatment. Questionnaire included 10 clinician-completed items. Each of 10 questions scored with a range of 0-6 points. An item score of 0 indicated item not present or normal, while an item score of 6 indicated severe or continuous presence of the symptoms. The total possible score was 60, and higher scores represented a more severe condition. A decrease in score by ≥ 50% indicated a response to treatment, and an actual score of ≤ 10 indicated a remission of symptoms.
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 38 | 34 | 38 | 37
units on a scale | -11.0 (11.59) | -12.7 (12.36) | -12.2 (10.50) | -17.3 (11.0) | -18.8 (10.33)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate) vs Arm 3- 50 μg MM-120 (LSD D-Tartrate) vs Arm 4- 100 μg MM-120 (LSD D-Tartrate) vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Assessment of change from baseline in total MADRS scores determined by the difference in means and difference between treatment and placebo (p-value determined from two-sample t-test); Test type: Superiority; p = 0.5538, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.6650, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0190, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0034, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores
Description: as for outcome 7
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 30 | 34 | 35 | 39 | 39
units on a scale | -12.4 (9.96) | -11.4 (11.63) | -12.3 (10.99) | -18.1 (11.97) | -18.3 (11.69)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Assessment of change from baseline in total CGI-S scores determined by the difference in means and difference between treatment and placebo (p-value determined from two-sample t-test); Test type: Superiority; p = 0.7236, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.9738, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0338, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0282, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores
Description: as for outcome 7
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 36 | 33
units on a scale | -12.2 (9.63) | -12.5 (11.88) | -11.1 (11.59) | -17.2 (12.66) | -18.6 (10.84)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.9302, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.6763, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0816, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0190, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Scores
Description: as for outcome 7
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale | -12.3 (9.53) | -13.9 (11.29) | -14.6 (8.57) | -18.7 (11.47) | -19.9 (11.15)
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.5647, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3497, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0229, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0073, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in anxiety symptoms measured via the CGI-S. The Clinical Global Impression - Severity (CGI-S) was used to assess the subject's current severity of illness at the time of the assessment relative to the clinician's past experience with patients who have the same diagnosis. The CGI-S comprises 1 Investigator-completed (or trained rater-completed) item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness. (minimum score 1, maximum score 7)
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 36
units on a scale
  change from Baseline | -1.0 [-1.46 to -0.54] | -1.8 [-2.18 to -1.34] | -1.7 [-2.20 to -1.19] | -2.3 [-2.67 to -1.85] | -2.4 [-2.80 to -1.97]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.76 [-1.38 to -0.15] | -0.69 [-1.37 to -0.02] | -1.26 [-1.87 to -0.66] | -1.39 [-2.00 to -0.78]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Change from baseline in total CGI-S scores determined by the difference in means and difference between treatment and placebo (p-value determined from two-sample t-test); Test type: Superiority; p = 0.0158, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0429, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0000, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Scores
Description: as for outcome 11
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 38 | 34 | 38 | 37
units on a scale
  change from baseline | -1.1 [-1.61 to -0.67] | -1.7 [-2.16 to -1.26] | -1.8 [-2.35 to -1.30] | -2.4 [-2.81 to -1.98] | -2.5 [-2.89 to -2.14]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.57 [-1.21 to 0.07] | -0.68 [-1.38 to 0.01] | -1.26 [-1.87 to -0.64] | -1.37 [-1.97 to -0.78]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0804, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0532, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0000, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Scores
Description: as for outcome 11
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 34 | 35 | 39 | 39
units on a scale
  Change from baseline | -1.3 [-1.85 to -0.79] | -1.8 [-2.25 to -1.28] | -1.7 [-2.12 to -1.19] | -2.5 [-2.93 to -2.05] | -2.3 [-2.74 to -1.88]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.44 [-1.15 to 0.26] | -0.33 [-1.03 to 0.36] | -1.16 [-1.84 to -0.49] | -0.99 [-1.65 to -0.32]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.2152, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3369, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0010, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0046, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Scores
Description: as for outcome 11
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Change from baseline | -1.5 [-2.15 to -0.88] | -1.8 [-2.28 to -1.34] | -1.7 [-2.18 to -1.13] | -2.3 [-2.74 to -1.83] | -2.5 [-2.99 to -2.04]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.29 [-1.07 to 0.48] | -0.14 [-0.94 to 0.67] | -0.77 [-1.53 to 0.00] | -1.00 [-1.77 to -0.22]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.4489, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.7326, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0492, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0131, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Scores
Description: as for outcome 11
Time Frame: End of Study (12 weeks)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale
  Change from baseline | -1.4 [-2.08 to -0.77] | -1.8 [-2.37 to -1.29] | -2.1 [-2.59 to -1.55] | -2.6 [-3.02 to -2.19] | -2.5 [-3.08 to -1.95]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.40 [-1.24 to 0.43] | -0.65 [-1.46 to 0.17] | -1.18 [-1.95 to -0.42] | -1.09 [-1.94 to -0.24]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.3330, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.1193, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0032, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0127, t-test, 2 sided

16. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in anxiety symptoms measured via the CGI-I. The Clinical Global Impression - Improvement (CGI-I) was used to measure the clinician's assessment of how much the subject's illness has improved or worsened relative to Baseline (Visit 2). The CGI-I comprises 1 Investigator-completed (or trained rater-completed) item with 7 possible ratings (1-7 points), where a lower score indicates improvement, and a higher score indicates worsening. (minimum score 1, maximum score 7)
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 35
units on a scale
  Actual Values CGI-I | 3.1 [2.69 to 3.49] | 2.4 [2.07 to 2.67] | 2.3 [1.98 to 2.69] | 1.8 [1.55 to 2.03] | 1.9 [1.61 to 2.16]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.72 [-1.21 to -0.23] | -0.75 [-1.28 to -0.23] | -1.30 [-1.76 to -0.84] | -1.20 [-1.68 to -0.73]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0046, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0052, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0000, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0000, t-test, 2 sided

17. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Total Scores
Description: as for outcome 16
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 38 | 34 | 38 | 37
units on a scale
  Actual values (CGI-I scores) | 3.0 [2.62 to 3.44] | 2.5 [2.13 to 2.87] | 2.4 [1.92 to 2.78] | 1.7 [1.43 to 1.94] | 1.9 [1.67 to 2.17]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.53 [-1.07 to 0.02] | -0.67 [-1.26 to -0.09] | -1.34 [-1.82 to -0.87] | -1.11 [-1.58 to -0.64]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0567, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0235, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0000, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0000, t-test, 2 sided

18. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Total Scores
Description: as for outcome 16
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 34 | 35 | 39 | 39
units on a scale
  Actual value (CGI-I score) | 2.8 [2.27 to 3.28] | 2.4 [2.00 to 2.82] | 2.4 [1.99 to 2.86] | 1.8 [1.51 to 2.08] | 2.2 [1.76 to 2.55]
  Difference in Means (MM120-placebo) | 0 [0 to 0] | -.036 [-1.00 to 0.28] | -0.35 [-1.00 to 0.31] | -0.98 [-1.56 to -0.40] | -0.62 [-1.25 to 0.01]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.2632, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.2962, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0013, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0547, t-test, 2 sided

19. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Total Scores
Description: as for outcome 16
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Actual vaues (CGI-I scores) | 2.7 [2.23 to 3.25] | 2.2 [1.86 to 2.58] | 2.7 [2.08 to 3.23] | 1.8 [1.51 to 2.15] | 2.0 [1.63 to 2.31]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.52 [-1.14 to 0.09] | -0.08 [-0.84 to 0.67] | -0.91 [-1.50 to -0.32] | -0.77 [-1.37 to -0.17]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0937, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.8230, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0032, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0129, t-test, 2 sided

20. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Total Scores
Description: as for outcome 16
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale
  Actual values (CGI-I scores) | 2.7 [2.19 to 3.27] | 2.3 [1.96 to 2.66] | 2.2 [1.68 to 2.73] | 1.6 [1.34 to 1.93] | 1.9 [1.46 to 2.35]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.42 [-1.06 to 0.21] | -0.52 [-1.26 to 0.21] | -1.09 [-1.70 to -0.49] | -0.83 [-1.52 to -0.14]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1889, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1589, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0008, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean CGI-I total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0194, t-test, 2 sided

21. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in anxiety symptoms measured via the PGI-S. The Patient Global Impression - Severity (PGI-S) is the patient-reported outcome counterpart to the CGI scale. The PGI is adapted to the patient population and can be used to measure disease severity (PGI-S). The PGI-S comprises 1 subject-completed item with 5 possible ratings (1-5). A higher score indicates more severe illness. (minimum score 1, maximum score 5)
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 36
units on a scale
  Change from baseline | -0.7 [-0.98 to -0.43] | -1.3 [-1.55 to -0.98] | -1.2 [-1.55 to -0.90] | -1.6 [-1.84 to -1.27] | -1.6 [-1.91 to -1.32]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.56 [-0.95 to -0.17] | -0.52 [-0.94 to -0.10] | -0.85 [-1.24 to -0.46] | -0.91 [-1.30 to -0.51]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Change from baseline in total PGI-S scores and the difference in means between treatment and placebo (p-value determined from two-sample t-test); Test type: Superiority; p = 0.0057, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0168, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Test type: Superiority; p = 0.0000, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0000, t-test, 2 sided

22. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Total Scores
Description: as for outcome 21
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 37 | 34 | 38 | 37
units on a scale
  Change from baseline | -0.8 [-1.10 to -0.45] | -1.2 [-1.49 to -0.83] | -1.3 [-1.65 to -0.88] | -1.5 [-1.80 to -1.15] | -1.6 [-1.88 to -1.26]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.38 [-0.84 to 0.07] | -0.49 [-0.98 to 0.01] | -0.70 [-1.15 to -0.25] | -0.79 [-1.23 to -0.35]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0958, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0544, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0029, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0006, t-test, 2 sided

23. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Total Scores
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 34 | 35 | 39 | 39
units on a scale
  Change from baseline | -1.0 [-1.35 to -0.65] | -1.3 [-1.70 to -0.95] | -1.3 [-1.66 to -0.97] | -1.5 [-1.78 to -1.19] | -1.6 [-1.94 to -1.19]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.32 [-0.83 to 0.18] | -0.31 [-0.80 to 0.17] | -0.49 [-0.94 to -0.03] | -0.56 [-1.07 to -0.06]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.2038, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.1977, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0357, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0302, t-test, 2 sided

24. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Total Scores
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Change from baseline | -1.0 [-1.41 to -0.52] | -1.3 [-1.67 to -0.95] | -1.1 [-1.58 to -0.61] | -1.4 [-1.70 to -1.05] | -1.6 [-2.05 to -1.22]
  difference in means (MM120-placebo) | 0 [0 to 0] | -0.35 [-0.91 to 0.21] | -0.13 [-0.78 to 0.52] | -0.41 [-0.95 to 0.13] | -0.67 [-1.27 to -0.08]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.2165, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.6868, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.1350, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.0273, t-test, 2 sided

25. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity (PGI-S) Total Scores
Description: as for outcome 21
Time Frame: End of study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale
  Change from baseline | -1.1 [-1.57 to -0.58] | -1.4 [-1.73 to -1.10] | -1.4 [-1.80 to -0.96] | -1.5 [-1.87 to -1.22] | -1.5 [-1.86 to -1.04]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.34 [-0.91 to 0.24] | -0.30 [-0.94 to 0.34] | -0.47 [-1.05 to 0.11] | -0.37 [-1.01 to 0.26]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.2450, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.3461, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.1110, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.2386, t-test, 2 sided

26. Secondary Outcome: Mean Patient Global Impression - Change (PGI-C) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in anxiety symptoms measured via the PGI-C. The Patient Global Impression - Change (PGI-C) is the patient-reported outcome counterpart to the CGI scale. The PGI is adapted to the patient population and can be used to measure changes in disease severity (PGI-C). The PGI-C comprises 1 subject-completed item with 5 possible ratings (1-5). A higher score indicates change for the worse (worsening symptoms). (minimum score 1, maximum score 5)
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 36
units on a scale
  Actual Values PGI-C | 2.3 [1.96 to 2.69] | 2.0 [1.74 to 2.26] | 1.8 [1.49 to 2.12] | 1.3 [1.14 to 1.55] | 1.5 [1.29 to 1.76]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.32 [-0.76 to 0.12] | -0.52 [-0.99 to -0.05] | -0.98 [-1.39 to -0.57] | -0.80 [-1.22 to -0.37]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1475, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0308, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0000, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0004, t-test, 2 sided

27. Secondary Outcome: Mean Patient Global Impression - Change (PGI-C) Total Scores
Description: as for outcome 26
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 37 | 34 | 38 | 37
units on a scale
  Actual values PGI-C | 2.4 [2.01 to 2.72] | 1.9 [1.61 to 2.28] | 2.0 [1.61 to 2.39] | 1.6 [1.31 to 1.85] | 1.5 [1.20 to 1.72]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.42 [-0.89 to 0.06] | -0.36 [-0.88 to 0.16] | -0.78 [-1.22 to -0.34] | -0.90 [-1.33 to -0.47]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0873, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1702, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0007, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0001, t-test, 2 sided

28. Secondary Outcome: Mean Patient Global Impression - Change (PGI-C) Total Scores
Description: as for outcome 26
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 34 | 35 | 39 | 39
units on a scale
  Actual values PGI-C | 2.3 [1.85 to 2.67] | 2.0 [1.63 to 2.43] | 1.9 [1.53 to 2.24] | 1.4 [1.17 to 1.55] | 1.7 [1.38 to 2.01]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.23 [-0.79 to 0.33] | -0.37 [-0.90 to 0.16] | -0.90 [-1.35 to -0.45] | -0.57 [-1.08 to -0.05]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.4193, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1663, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0002, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0306, t-test, 2 sided

29. Secondary Outcome: Mean Patient Global Impression - Change (PGI-C) Total Scores
Description: as for outcome 26
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Actual values PGI-C | 2.1 [1.79 to 2.51] | 1.7 [1.46 to 1.98] | 2.0 [1.64 to 2.42] | 1.5 [1.27 to 1.81] | 1.8 [1.41 to 2.10]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.43 [-0.87 to 0.01] | -0.12 [-0.64 to 0.40] | -0.61 [-1.04 to -0.17] | -0.39 [-0.88 to 0.10]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0534, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.6551, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0079, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1133, t-test, 2 sided

30. Secondary Outcome: Change From Baseline in Patient Global Impression - Change (PGI-C) Total Scores
Description: as for outcome 26
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale
  Actual values PGI-C | 2.2 [1.80 to 2.59] | 1.8 [1.56 to 2.10] | 1.8 [1.45 to 2.21] | 1.5 [1.25 to 1.72] | 1.7 [1.32 to 2.04]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.36 [-0.83 to 0.10] | -0.36 [-0.90 to 0.17] | -0.71 [-1.16 to -0.25] | -0.51 [-1.04 to 0.01]
Statistical Analysis 1: Comparison: Arm 1- Placebo vs Arm 2- 25 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1248, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm 1- Placebo vs Arm 3- 50 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.1788, t-test, 2 sided
Statistical Analysis 3: Comparison: Arm 1- Placebo vs Arm 4- 100 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0030, t-test, 2 sided
Statistical Analysis 4: Comparison: Arm 1- Placebo vs Arm 5- 200 μg MM-120 (LSD D-Tartrate); Difference in mean PGI-C total scores (MM120-placebo); p-value determined from two-sample t-test; Test type: Superiority; p = 0.0534, t-test, 2 sided

31. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Scores
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in functional disability symptoms measured via the SDS. The Sheehan Disability Scale (SDS) is a composite of 3 self-rated items designed to measure the extent to which 3 major domains in the patient's life (work, social life/leisure activities and family life/home responsibilities) are functionally impaired by psychiatric or medical symptoms. Total score 0-30 (0 unimpaired, 30 highly impaired). Work/school (0-10); Social life (0-10); Family life/home responsibilities (0-10).
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 35
units on a scale
  Change from baseline | -7.4 [-10.00 to -4.83] | -8.8 [-10.91 to -6.67] | -8.0 [-10.73 to -5.33] | -14.6 [-16.67 to -12.49] | -13.6 [-15.61 to -11.59]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.38 [-4.66 to 1.91] | -0.62 [-4.29 to 3.05] | -7.17 [-10.44 to -3.90] | -6.19 [-9.40 to -2.97]

32. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Scores
Description: as for outcome 31
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 37 | 34 | 38 | 36
units on a scale
  Change from Baseline | -7.8 [-10.49 to -5.18] | -9.8 [-12.32 to -7.30] | -8.2 [-11.04 to -5.43] | -14.0 [-16.23 to -11.71] | -14.2 [-16.42 to -11.97]
  Difference in means (MM120-placeb) | 0 [0 to 0] | -1.98 [-5.57 to 1.61] | -0.40 [-4.20 to 3.39] | -6.14 [-9.57 to -2.71] | -6.36 [-9.77 to -2.95]

33. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Scores
Description: as for outcome 31
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 33 | 34 | 39 | 39
units on a scale
  Change from baseline | -9.0 [-12.03 to -5.90] | -9.5 [-12.24 to -6.67] | -8.7 [-11.41 to -5.94] | -14.9 [-17.18 to -12.66] | -13.5 [-15.88 to -11.04]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.49 [-4.55 to 3.58] | 0.29 [-3.74 to 4.32] | -5.96 [-9.70 to -2.21] | -4.49 [-8.33 to -0.66]

34. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Scores
Description: as for outcome 31
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Change from baseline | -9.1 [-12.62 to -5.68] | -10.5 [-13.21 to -7.73] | -7.5 [-10.77 to -4.17] | -13.8 [-16.48 to -11.18] | -13.6 [-16.39 to -10.76]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.32 [-5.65 to 3.01] | 1.68 [-3.01 to 6.37] | -4.68 [-8.96 to -0.40] | -4.43 [-8.81 to -0.05]

35. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Scores
Description: as for outcome 31
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 25 | 29 | 29 | 33 | 31
units on a scale
  Change from baseline | -8.2 [-11.75 to -4.65] | -10.8 [-13.73 to -7.85] | -9.0 [-12.52 to -5.54] | -15.1 [-17.11 to -13.01] | -13.1 [-15.88 to -10.37]
  Difference in means (MM120-plcebo) | 0 [0 to 0] | -2.59 [-7.10 to 1.91] | -0.83 [-5.70 to 4.03] | -6.86 [-10.89 to -2.83] | -4.93 [-9.33 to -0.53]

36. Secondary Outcome: Improved Quality of Life as Measured by EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in quality of life. The EuroQol 5 Dimension 5 Level (EQ-5D-5L) was used to evaluate health outcomes over a wide range of health conditions and treatments. The EQ-5D consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The VAS for the subject's health status scored as ranging from 0 = worst health you can imagine, to 100 = best health you can imagine.
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 34 | 38 | 36 | 38 | 36
units on a scale
  Change from baseline | 6.9 [1.08 to 12.69] | 11.2 [4.57 to 17.85] | 12.3 [7.15 to 17.46] | 15.7 [10.20 to 21.12] | 14.9 [9.79 to 19.93]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 4.33 [-4.34 to 13.00] | 5.43 [-2.20 to 13.05] | 8.78 [0.95 to 16.60] | 7.98 [0.41 to 15.55]

37. Secondary Outcome: Improved Quality of Life as Measured by EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: as for outcome 36
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 36 | 37 | 34 | 38 | 37
units on a scale
  Change from baseline | 10.3 [5.49 to 15.12] | 11.8 [4.66 to 18.85] | 10.6 [5.51 to 15.61] | 14.7 [9.72 to 19.64] | 15.9 [10.46 to 21.27]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 1.45 [-6.99 to 9.89] | 0.25 [-6.60 to 7.10] | 4.38 [-2.41 to 11.17] | 5.56 [-1.55 to 12.67]

38. Secondary Outcome: Improved Quality of Life as Measured by EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: as for outcome 36
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 31 | 33 | 35 | 38 | 39
units on a scale
  Change from baseline | 11.5 [5.79 to 17.17] | 13.5 [5.76 to 21.33] | 10.5 [4.76 to 16.33] | 15.5 [10.27 to 20.73] | 15.7 [9.02 to 22.32]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 2.03 [-7.41 to 11.53] | -0.94 [-8.90 to 7.02] | 4.02 [-3.57 to 11.60] | 4.18 [-4.41 to 12.78]

39. Secondary Outcome: Improved Quality of Life as Measured by EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 32 | 32 | 35 | 33
units on a scale
  Change from baseline | 10.8 [3.97 to 17.66] | 16.2 [10.20 to 22.18] | 9.7 [3.37 to 16.07] | 16.2 [9.94 to 22.52] | 17.0 [10.07 to 23.93]
  Diference in means (MM120-placebo) | 0 [0 to 0] | 5.37 [-3.53 to 14.28] | -1.10 [-10.23 to 8.04] | 5.41 [-3.69 to 14.52] | 6.19 [-3.35 to 15.72]

40. Secondary Outcome: Improved Quality of Life as Measured by EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: as for outcome 36
Time Frame: End of Study (12 weeks)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 29 | 33 | 31
units on a scale
  Change from baseline | 11.7 [4.28 to 19.02] | 17.0 [9.92 to 24.01] | 13.2 [7.89 to 18.52] | 17.7 [12.85 to 22.55] | 17.3 [10.18 to 24.40]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 5.31 [-4.65 to 15.27] | 1.55 [-7.34 to 10.45] | 6.04 [-2.61 to 14.70] | 5.64 [-4.37 to 15.65]

41. Secondary Outcome: Improved Sleep as Measured by Pittsburgh Sleep Quality Index (PSQI)
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in subjects with anxiety symptoms, including improvements in sleep measured via the PSQI. The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality and disturbances over the preceding month. The questionnaire had a Component Score for each of these with a range of 0-3 points: Subjective sleep quality, Sleep latency, Sleep duration, Habitual sleep efficiency, Sleep disturbance, Use of sleeping medication, and Daytime dysfunction. The sum of the Component Scores = a Global Score. Global Score of 0 indicated no difficulty and a Global Score of 21 indicated severe difficulty in all areas.
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 32 | 37 | 33 | 38 | 39
units on a scale
  Change from baseline | -3.7 [-5.10 to -2.21] | -3.8 [-5.20 to -2.37] | -2.7 [-4.32 to -1.14] | -5.3 [-6.57 to -4.01] | -3.9 [-5.04 to -2.75]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.13 [-2.11 to 1.86] | 0.93 [-1.18 to 3.04] | -1.63 [-3.53 to 0.26] | -0.24 [-2.05 to 1.57]

42. Secondary Outcome: Improved Sleep as Measured by Pittsburgh Sleep Quality Index (PSQI)
Description: as for outcome 41
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 27 | 31 | 32 | 35 | 32
units on a scale
  Change from baseline | -4.1 [-5.70 to -2.60] | -5.4 [-6.97 to -3.80] | -3.6 [-5.21 to -1.98] | -5.1 [-6.61 to -3.67] | -4.4 [-5.94 to -2.88]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.24 [-3.41 to 0.93] | 0.55 [-1.63 to 2.74] | -0.99 [-3.09 to 1.10] | -0.26 [-2.39 to 1.87]

43. Secondary Outcome: Improved Sleep as Measured by Pittsburgh Sleep Quality Index (PSQI)
Description: as for outcome 41
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 26 | 29 | 28 | 33 | 31
units on a scale
  Change from baseline | -4.3 [-5.97 to -2.56] | -5.5 [-7.04 to -3.99] | -4.8 [-6.33 to -3.32] | -5.9 [-7.37 to -4.45] | -4.9 [-6.38 to -3.36]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.25 [-3.48 to 0.99] | -0.55 [-2.77 to 1.67] | -1.64 [-3.84 to 0.56] | -0.60 [-2.83 to 1.62]

44. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Females
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in female subjects with anxiety symptoms, including improvements in sexual function measured via the ASEX. The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction.
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 23 | 20 | 20 | 16 | 24
units on a scale
  Change from baseline | -2.1 [-4.46 to 0.20] | -1.4 [-3.70 to 0.90] | -1.9 [-3.54 to -0.16] | -3.1 [-5.56 to -0.58] | -2.5 [-4.35 to -0.73]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 0.73 [-2.44 to 3.90] | 0.28 [-2.52 to 3.08] | -0.94 [-4.22 to 2.35] | -0.41 [-3.29 to 2.46]

45. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Females
Description: as for outcome 44
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 25 | 20 | 19 | 14 | 27
units on a scale
  Change from baseline | -1.0 [-2.83 to 0.83] | -2.2 [-4.07 to -0.33] | 0.4 [-1.33 to 2.18] | -2.4 [-4.70 to -0.02] | -2.2 [-4.10 to -0.34]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.20 [-3.74 to 1.34] | 1.42 [-1.04 to 3.88] | -1.36 [-4.22 to 1.50] | -1.22 [-3.78 to 1.34]

46. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Females
Description: as for outcome 44
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 21 | 18 | 19 | 16 | 28
units on a scale
  Change from Baseline | -3.6 [-6.07 to -1.17] | -2.5 [-3.99 to -1.01] | -1.1 [-2.72 to 0.51] | -3.3 [-5.76 to -0.77] | -1.2 [-3.17 to 0.81]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 1.12 [-1.67 to 3.91] | 2.51 [-0.34 to 5.37] | 0.35 [-3.01 to 3.72] | 2.44 [-0.63 to 5.51]

47. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Females
Description: as for outcome 44
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 19 | 17 | 17 | 14 | 24
units on a scale
  Change from baseline | -4.4 [-7.33 to -1.51] | -2.0 [-3.74 to -0.26] | -0.7 [-2.29 to 0.88] | -1.8 [-4.19 to 0.65] | -2.8 [-4.38 to -1.20]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 2.42 [-0.87 to 5.71] | 3.72 [0.49 to 6.94] | 2.65 [-0.97 to 6.27] | 1.63 [-1.61 to 4.87]

48. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Females
Description: as for outcome 44
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 18 | 16 | 15 | 13 | 21
units on a scale
  Change from baseline | -3.9 [-6.77 to -1.12] | -2.7 [-4.83 to -0.55] | -1.3 [-3.56 to 0.90] | -2.8 [-5.45 to -0.09] | -2.7 [-4.38 to -1.05]
  Difference in means (MM120-placebo) | 0 [0 to 0] | 1.26 [-2.15 to 4.67] | 2.61 [-0.85 to 6.07] | 1.18 [-2.54 to 4.89] | 1.23 [-1.96 to 4.42]

49. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Males
Description: To determine whether MM120 (25, 50, 100, or 200 µg freebase-equivalent) improves functionality and quality of life measures in male subjects with anxiety symptoms, including improvements in sexual function measured via the ASEX. The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction.
Time Frame: Week 1
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 10 | 18 | 16 | 22 | 12
units on a scale
  Change from baseline | 0.1 [-1.88 to 2.08] | -1.4 [-2.57 to -0.21] | -0.6 [-2.88 to 1.63] | -1.1 [-2.90 to 0.63] | -1.1 [-3.41 to 1.24]
  Difference in mean (MM120-placebo) | 0 [0 to 0] | -1.49 [-3.69 to 0.71] | -0.73 [-3.56 to 2.11] | -1.24 [-3.75 to 1.28] | -1.18 [-4.04 to 1.68]

50. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Males
Description: as for outcome 49
Time Frame: Week 2
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 11 | 17 | 15 | 24 | 10
units on a scale
  Change from baseline | 0.0 [-2.23 to 2.23] | -1.1 [-2.51 to 0.28] | -0.5 [-3.06 to 2.13] | -1.3 [-2.71 to 0.21] | -0.6 [-2.39 to 1.19]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.12 [-3.63 to 1.39] | -0.47 [-3.71 to 2.77] | -1.25 [-3.80 to 1.30] | -0.60 [-3.28 to 2.08]

51. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Males
Description: as for outcome 49
Time Frame: Week 4
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 10 | 15 | 16 | 23 | 11
units on a scale
  Change from baseline | -0.2 [-2.53 to 2.13] | -1.3 [-3.17 to 0.50] | -0.9 [-3.02 to 1.27] | -2.1 [-3.97 to -0.29] | -1.6 [-5.33 to 2.06]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.13 [-3.93 to 1.66] | -0.68 [-3.66 to 2.31] | -1.93 [-4.75 to 0.89] | -1.44 [-5.57 to 2.69]

52. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Males
Description: as for outcome 49
Time Frame: Week 8
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 8 | 14 | 15 | 21 | 9
units on a scale
  Change from baseline | -1.1 [-6.05 to 3.80] | -1.3 [-3.46 to 0.89] | -1.4 [-3.07 to 0.27] | -2.0 [-3.47 to -0.43] | -3.2 [-8.19 to 1.74]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -0.16 [-5.29 to 4.97] | -0.28 [-5.30 to 4.75] | -0.83 [-5.84 to 4.18] | -2.10 [-8.48 to 4.29]

53. Secondary Outcome: Improved Sexual Functioning as Measured by Arizona Sexual Experiences Questionnaire (ASEX) - Males
Description: as for outcome 49
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 8 | 13 | 14 | 20 | 10
units on a scale
  Change from baseline | -0.3 [-2.73 to 2.23] | -1.3 [-2.93 to 0.32] | -2.4 [-3.86 to -1.00] | -1.9 [-3.21 to -0.59] | -2.5 [-6.35 to 1.35]
  Difference in means (MM120-placebo) | 0 [0 to 0] | -1.06 [-3.82 to 1.70] | -2.18 [-4.86 to 0.51] | -1.65 [-4.30 to 1.00] | -2.25 [-6.52 to 2.02]

54. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Females, to Week 1
Description: Number of Participants with sexual dysfunction n (%) vs Number of Participants without sexual dysfunction n (%). The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction.
Time Frame: Week 1
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 23 | 20 | 20 | 16 | 24
Participants
  Number of Participants with sexual dysfunction | 12 | 10 | 9 | 6 | 8
  Number of Participants without sexual dysfunction | 11 | 10 | 11 | 10 | 16

55. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Females, to Week 2
Description: as for outcome 54
Time Frame: Week 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 25 | 20 | 19 | 14 | 27
Participants
  Number of Participants with sexual dysfunction | 14 | 7 | 14 | 5 | 10
  Number of Participants without sexual dysfunction | 11 | 13 | 5 | 9 | 17

56. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Females, to Week 4
Description: as for outcome 54
Time Frame: Week 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 21 | 19 | 19 | 16 | 28
Participants
  Number of Participants with sexual dysfunction | 8 | 6 | 11 | 6 | 10
  Number of Participants without sexual dysfunction | 13 | 13 | 8 | 10 | 18

57. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Females, to Week 8
Description: Number of Participants with sexual dysfunction n (%) vs. Number of Participants without sexual dysfunction n (%). The Arizona Sexual Experiences Questionnaire (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm over the past week. Possible total scores on the ASEX range of 5-30, with a higher score indicating more sexual dysfunction.
Time Frame: Week 8
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 19 | 17 | 17 | 14 | 24
Participants
  Number of Participants with sexual dysfunction | 5 | 6 | 11 | 6 | 8
  Number of Participants without sexual dysfunction | 14 | 11 | 6 | 8 | 16

58. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Females, to Week 12
Description: as for outcome 57
Time Frame: End of Study (Week 12)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 18 | 16 | 15 | 13 | 21
Participants
  Number of Participants with sexual dysfunction | 6 | 4 | 10 | 6 | 7
  Number of Participants without sexual dysfunction | 12 | 12 | 5 | 7 | 14

59. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Males, to Week 1
Description: as for outcome 57
Time Frame: Week 1
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 10 | 18 | 16 | 22 | 12
Participants
  Number of Participants with sexual dysfunction | 1 | 4 | 3 | 2 | 3
  Number of Participants without sexual dysfunction | 9 | 14 | 13 | 20 | 9

60. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Males, to Week 2
Description: as for outcome 57
Time Frame: Week 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 11 | 17 | 15 | 24 | 10
Participants
  Number of Participants with sexual dysfunction | 0 | 3 | 3 | 2 | 1
  Number of Participants without sexual dysfunction | 11 | 14 | 12 | 22 | 9

61. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Males, to Week 4
Description: as for outcome 57
Time Frame: Week 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 10 | 15 | 16 | 23 | 11
Participants
  Number of Participants with sexual dysfunction | 0 | 3 | 4 | 1 | 0
  Number of Participants without sexual dysfunction | 10 | 12 | 12 | 22 | 11

62. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Males, to Week 8
Description: as for outcome 57
Time Frame: Week 8
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 8 | 15 | 15 | 21 | 9
Participants
  Number of Participants with sexual dysfunction | 1 | 3 | 4 | 1 | 1
  Number of Participants without sexual dysfunction | 7 | 12 | 11 | 20 | 8

63. Secondary Outcome: Summary of Sexual Dysfunction Rates (ASEX), Males, to Week 12
Description: as for outcome 57
Time Frame: Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
Number analyzed (Participants) | 8 | 13 | 14 | 20 | 10
Participants
  Number of Participants with sexual dysfunction | 1 | 3 | 1 | 2 | 0
  Number of Participants without sexual dysfunction | 7 | 10 | 13 | 18 | 10

ADVERSE EVENTS:
Time Frame: AE collection will occur from the time informed consent is given until Week 12 (or early discontinuation) and will be recorded at each visit.
Arm/Group | Arm 1- Placebo | Arm 2- 25 μg MM-120 (LSD D-Tartrate) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) | Arm 5- 200 μg MM-120 (LSD D-Tartrate)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 1/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 22/39 | 30/39 | 36/40 | 39/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- Placebo (N=39) | Arm 2- 25 μg MM-120 (LSD D-Tartrate) (N=39) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) (N=40) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) (N=40) | Arm 5- 200 μg MM-120 (LSD D-Tartrate) (N=40)
Panic Attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 — Participant received MM120 on 26 January 2023. On Study Day 98, the participant experienced an SAE of moderate panic attack requiring hospitalization. It was considered not related to treatment and recovered same day.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Placebo (N=39) | Arm 2- 25 μg MM-120 (LSD D-Tartrate) (N=39) | Arm 3- 50 μg MM-120 (LSD D-Tartrate) (N=40) | Arm 4- 100 μg MM-120 (LSD D-Tartrate) (N=40) | Arm 5- 200 μg MM-120 (LSD D-Tartrate) (N=40)
Illusion (Psychiatric disorders) | 3 (3) | 12 (15) | 18 (23) | 25 (31) | 30 (46)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (5) | 11 (12) | 16 (21) | 24 (31)
Headaches (Nervous system disorders) | 9 (12) | 5 (6) | 9 (11) | 14 (16) | 11 (13)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 6 (7) | 9 (10) | 9 (10) | 6 (6)
Euphoric mood (Psychiatric disorders) | 1 (1) | 2 (2) | 5 (6) | 11 (11) | 6 (8)
Amxiety (Psychiatric disorders) | 2 (2) | 4 (4) | 5 (6) | 4 (4) | 6 (7)
Mydriasis (Eye disorders) | 1 (1) | 1 (1) | 7 (7) | 8 (8) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 9 (9) | 5 (5)
Fatigue (General disorders) | 1 (1) | 2 (2) | 6 (8) | 4 (4) | 4 (4)
Blood pressure increased (Investigations) | 0 (0) | 3 (3) | 5 (5) | 4 (5) | 4 (4)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 8 (8)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (5) | 4 (4) | 4 (7)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 5 (5)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 5 (6) | 5 (5)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 8 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 5 (6)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (8) | 0 (0) | 1 (1)
Pseudohallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Feeling abnormal (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Tearfulness (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Derealisation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Heart rate increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Feeling drunk (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Irritabilty (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0)
Time percetion altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Depersonalisation/derealisation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Feeling of relaxation (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pollakuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Autoscopy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Inappropriate affect (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Logorrhoea (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Motor dysfunction (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
DSMs assisted and monitored participants which could be construed to have an independent therapeutic effect. So, DSMs were given training to not engage in psychotherapy with participants.

There was a potential for unblinding so blinded independent central raters assessed the primary efficacy outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Sponsor has at least 60 days to review a proposed publication before submission for purposes of requesting the removal of Sponsor's confidential information.
2. Institutions and PI's will not publish or disclosure their single-site data prior to a multi-center publication of the aggregate study data, unless Sponsor does not publish a multi-center publication within 12 months following conclusion of the overall study.

DOCUMENTS (2):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT05407064/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT05407064/SAP_002.pdf